CLINICAL TRIAL: NCT03162276
Title: Evaluating the Effectiveness of Inquiry Based Stress Reduction (IBSR) Intervention Versus Regular Care of no Treatment on Well-being, Optimism and Health Behavior of BRCA1/2 Carriers: A Randomized Controlled Trial, RCT.
Brief Title: Trial of Inquiry Based Stress Reduction (IBSR) Program for BRCA1/2 Mutation Carriers
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-17-3856-EF-CTIL
Record Dates: First submitted 2017-05-07; First posted 2017-05-22 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome
Keywords: BRCA 1/2 Carriers; The Work; RCT; IBSR
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Inquiry Based Stress Reduction
  Interventions: Behavioral: Inquiry Based Stress Reduction (IBSR) program
- Control (Placebo Comparator): The placebo group participants will receive a modified form of the intervention at the close of the study
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Inquiry Based Stress Reduction (IBSR) program — The IBSR (Inquiry-based stress reduction) intervention, developed by Byron Katie, trains participants to reduce their perceived level of stress by self-inquiry of their thoughts and beliefs connected to stressful circumstances or symptoms. This meditative process, named "The Work", enables the participants to identify and question the stressful thoughts that cause their suffering. The core of IBSR is simply four questions and a turnaround, which is a way of experiencing the opposite of what the participant believes. This process is simple, powerful and provides skills for self-inquiry and management of stressful thoughts that can be easily implemented in daily life
  Arms: Intervention
Behavioral: Control — At end of intervention, the control group will receive a brief intervention consisting of a home kit for practicing IBSR techniques.
  Arms: Control

SUMMARY:
Breast cancer (BC) is a major health problem and the most prevalent cancer among women.In a substantial proportion of familial cases, germ-line mutations in either BRCA1/2 can be detected. The only proven modality for active risk reduction (rather than passive early detection), is prophylactic surgery - prophylactic mastectomy and oophorectomy. While the majority of Jewish mutation carriers elect to undergo prophylactic oophorectomy at about age 40 years, in Israel only a minority perform prophylactic mastectomy. Another ramification of being a mutation carrier is the emotional stress associated with that discovery.Genetic information has profound implications for mutation carriers. The IBSR (Inquiry-based stress reduction) intervention, developed by Byron Katie, trains participants to reduce their perceived level of stress by self-inquiry of their thoughts and beliefs connected to stressful circumstances or symptoms. This meditative process, named "The Work", enables the participants to identify and question the stressful thoughts that cause their suffering. The core of IBSR is simply four questions and a turnaround, which is a way of experiencing the opposite of what the participant believes. This process is simple, powerful and provides skills for self-inquiry and management of stressful thoughts that can be easily implemented in daily life [ ]. Therefore, on the basis of previous data and beneficial observations we postulate that the clinical utility of IBSR mediation program may improve psychological and physical symptoms and quality of life among asymptomatic (oncologically healthy) BRCA1/ BRCA2 mutation carriers. Thus, we will conduct a pilot randomized controlled trial to scientifically investigate the effect of this intervention effects on BRCA1/2 mutation carriers.

DETAILED DESCRIPTION:
Primary goal: to evaluate the effectiveness of IBSR intervention on psychological well-being of BRCA carriers.

Secondary goals:

* To understand the IBSR action mechanism and to develop a theoretical model.
* To examine the correlation between psychological well-being and optimism and health behaviors among carriers.
* To evaluate and define core beliefs related to psychological well-being, optimism and expectations among carriers.
* To evaluate and define the health related behaviors among carriers.

Rationale for studies: The rationale of the research emerges from two aspects. One aspect is the effort to establish a new intervention program for women in order to help them deal with the daily implications of being a BRCA carrier. Up to date, only few interventions were carried out in Israel and worldwide, and had several methodological limitations.

The other aspect is the combination of quantitative and qualitative tools in order to analyze the psychological implications of a complicated medical state and to establish an intervention program in order to reduce their adverse impact. This combination can significantly contribute to the understanding of the investigated issue and the participants' experience. The current research is comprehensive and rigorous, and it is based on a randomized controlled study, which was carried out with 118 Israeli women.

Research plan and milestones:

Research Design: A randomized controlled study offering IBSR intervention for BRCA carriers.

Research sample: 118 asymptomatic BRCA1/2 carriers, being followed-up in the high-risk clinic at Sheba hospital and meet the inclusion criteria:

asymptomatic carriers of BRCA1/2 mutation, level of Hebrew, age group and psychiatric illness. Age: 25-55

Intervention group: 59 carriers who will participate in a 8-12 sessions (up to 48 hours) group workshop of IBSR.

Control group: 59 carriers who will not participate in the workshop. They will complete questionnaires on the same time points as the intervention group. Participants who completed all the questionnaires will receive an IBSR kit for home practice.

Research outcomes: psychological well-being, optimism, satisfaction with life, mental well-being, quality of sleep health behaviors and perceptions. In addition, the main themes from the qualitative interviews.

ELIGIBILITY:
Inclusion Criteria:

* Women who are carriers of one of the predominant Jewish mutations in BRCA1/2 genes, age 25-55 years, with no current or past history of cancer (except BCC), who are willing to sign an informed consent, and present mental clarity by the ability to comprehend and fulfill all the questionnaires.

Exclusion Criteria:

* Diagnosed with breast or ovarian cancer or any other cancer, risk reduction mastectomy, severe psychiatric diagnosis (e.g. bipolar disorder).

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
The Ryff scale- Psychological well-being | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  Questionnaire

SECONDARY OUTCOMES:
Life Orientation Test-Revise- LOT-R | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire assesses the degree of optimism
Satisfaction with life scale - SWLS d | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire assesses the degree of Satisfaction with the life
Pittsburgh Sleep Quality Inventory Questionnaire- PSQI | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire assesses the quality of sleep
Positive and negative affect schedule PANAS | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire assesses the degree of positive and negative feelings
Self-assessed health SAH | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire assesses the personal perceived health
Euroqol quality of life scale EQ-5D | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire assesses the quality of life
Perceived social support from family PSS-FA | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire assesses the perceived family support
Mindfulness attention awareness scale MAAS | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire assesses the degree of mindfulness attention
General self- efficacy GSE | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire assesses the degree of self- efficacy
Demographic and behavioral data | A measure assessing change between 3 time points (before the intervention, after 5 months (at the end of the intervention) and 3 months later)
  This questionnaire asks about demographics data and health behavior

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Friedman, Prof., Principal Investigator — Sheba Medical Center; Carla Landau, Ph.D Student, Principal Investigator — Tel Aviv University; Shahar Lev- Ari, Dr., Principal Investigator — Tel Aviv University; Laura Rosen, Dr., Principal Investigator — Tel Aviv University
Locations (2):
- Israel (2):
  - Sheba Medical Center, Tel Aviv
  - Eitan Friedman, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Landau C, Lev-Ari S, Cohen-Mansfield J, Tillinger E, Geva R, Tarrasch R, Mitnik I, Friedman E. Randomized controlled trial of Inquiry-Based Stress Reduction (IBSR) technique for BRCA1/2 mutation carriers. Psychooncology. 2015 Jun;24(6):726-31. doi: 10.1002/pon.3703. Epub 2014 Oct 18. No abstract available. PMID 25328041
- [Background] Landau C, Mitnik I, Cohen-Mensfild J, Tillinger E, Geva R, , Friedman E. Lev-Ari S. Inquiry-based stress reduction (IBSR) meditation technique for brCA1/2 mutation carriers-A qualitative study. European Journal of Integrative Medicine; Dec 2016; 8 (6): 958-964
- [Derived] Landau C, Novak AM, Ganz AB, Rolnik B, Friedman E, Lev-Ari S. Effect of Inquiry-Based Stress Reduction on Well-being and Views on Risk-Reducing Surgery Among Women With BRCA Variants in Israel: A Randomized Clinical Trial. JAMA Netw Open. 2021 Dec 1;4(12):e2139670. doi: 10.1001/jamanetworkopen.2021.39670. PMID 34962562